CLINICAL TRIAL: NCT00237003
Title: A Brief Alcohol Intervention for Incarcerated Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Michael Stein, MD, Butler Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIAAASTE14495; R01AA014495 (NIH); NIAAASTE14495
Record Dates: First submitted 2005-10-11; First posted 2005-10-12 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-05

CONDITIONS: Alcohol Use; Incarceration
Keywords: women; incarceration; alcohol use; motivational interviewing
MeSH Terms: conditions — Alcohol Drinking | interventions — Motivational Interviewing

ARMS (1):
- 1) assessment plus motivational interview (Active Comparator): Participants are assigned, in this 6 month study, to an assessment-only condition or an assessment plus motivational interview condition. Two motivational interview sessions are conducted during the first month of study participation.
  Interventions: Behavioral: motivational interviewing

INTERVENTIONS:
Behavioral: motivational interviewing — Assessment plus motivational interview condition -- two motivational interview sessions are conducted during the first month of this six month study participation.

SUMMARY:
The purpose of this study is to examine the efficacy of a brief motivational intervention for alcohol use in incarcerated women.

DETAILED DESCRIPTION:
Hazardous alcohol use continues to be a problem of major significance throughout the United States. Alcohol use is a prevalent condition that independently acts as an important behavioral cofactor for HIV infection in women, contributing to both sexual and drug risk. The rationale for a brief intervention with incarcerated women who hazardously use alcohol and have HIV risk behaviors is compelling. For such women, we believe that the negative effects of drinking may be increased. An intervention that successfully connects alcohol use with HIV risk behaviors may be sufficient to tip the decisional balance in favor of reducing risk-prone alcohol consumption. If alcohol consumption is reduced more generally in a person's life, this may improve judgment in pursuing behaviors which risk other negative consequences. Hazardous alcohol, and high-risk drug and sexual activities may be manifestations of a general behavior pattern among incarcerated women, and strategies that engage such individuals are needed. Given the strong association between hazardous alcohol use and high HIV risk sexual and drug activities, interventions that attempt to lower the prevalence of HIV drug and sexual risk activities by lowering alcohol consumption are well justified. Brief alcohol interventions have been efficacious in reducing alcohol use across many populations over the past decade.

Comparison(s): Participants are assigned, in this 6 month study, to an assessment-only condition or an assessment plus motivational interview condition. Two motivational interview sessions are conducted during the first month of study participation.

ELIGIBILITY:
Inclusion Criteria:

* incarcerated women
* current hazardous drinking
* current HIV risk behavior

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Estimated)
Dates: Start 2003-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
alcohol use | 6 months
HIV risk taking | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stein, M.D., Principal Investigator — Butler Hospital

REFERENCES:
- [Derived] Hayaki J, Anderson BJ, Stein MD. Sexual risk-taking mediates the association between impulsivity and acquisition of sexually transmitted infections among hazardously drinking incarcerated women. Am J Addict. 2012 Nov;21 Suppl 1(Suppl 1):S63-71. doi: 10.1111/j.1521-0391.2012.00296.x. PMID 23786513
- [Derived] Caviness CM, Anderson BJ, de Dios MA, Kurth M, Stein M. Prescription medication exchange patterns among methadone maintenance patients. Drug Alcohol Depend. 2013 Jan 1;127(1-3):232-8. doi: 10.1016/j.drugalcdep.2012.07.007. Epub 2012 Jul 31. PMID 22854293
- [Derived] Caviness CM, Anderson BJ, Stein MD. Prevalence and predictors of sexually transmitted infections in hazardously-drinking incarcerated women. Women Health. 2012;52(2):119-34. doi: 10.1080/03630242.2011.649396. PMID 22458289
- [Derived] Clarke JG, Anderson BJ, Stein MD. Hazardously drinking women leaving jail: time to first drink. J Correct Health Care. 2011 Jan;17(1):61-8. doi: 10.1177/1078345810385915. PMID 21278321
- [Derived] Stein MD, Caviness CM, Anderson BJ, Hebert M, Clarke JG. A brief alcohol intervention for hazardously drinking incarcerated women. Addiction. 2010 Mar;105(3):466-75. doi: 10.1111/j.1360-0443.2009.02813.x. PMID 20402990
- [Derived] Stein MD, Anderson BJ, Caviness CM, Rosengard C, Kiene S, Friedmann P, Clarke JG. Relationship of alcohol use and sexual risk taking among hazardously drinking incarcerated women: an event-level analysis. J Stud Alcohol Drugs. 2009 Jul;70(4):508-15. doi: 10.15288/jsad.2009.70.508. PMID 19515290